CLINICAL TRIAL: NCT00855829
Title: A Single-Center, Randomized, Controlled, Double-Blind Feasibility Study Designed to Assess the Safety Performance of ActiLady Prototype in Adult Female Subjects With Dysmenorrhea.
Brief Title: A Feasibility Study Designed to Assess the Efficacy of the ActiLady Device in Adult Female Subjects With Dysmenorrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ezra Yosi, Prof. Yossi Ezra, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: galmedics-HMO-CTIL
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miniature Actilady device active (Active Comparator): one miniature Actilady device tested for all patients during a 4 months period. The device is active in 3 months out of the 4, and the patients are blinded to the action of the device (sham comparator).
  Interventions: Device: Miniature Actilady device active
- Miniature Actilady device not active (Sham Comparator): Sham Comparator: one miniature Actilady device tested for all patients during a 4 months period. The device is active in 3 months out of the 4, and the patients are blinded to the action of the device (sham comparator).
  Interventions: Device: Miniature Actilady device not active

INTERVENTIONS:
Device: Miniature Actilady device active — Devices: Targeted pressure waves are created by two kind of methods ActiLady).
  1. The effect of the waves used will be examined by the use of a silicon tube or polyvinyl chloride (PVC) tube which is inserted into the vaginal cavity. The other end of the tube will be connected to an "off the shelf" pressure waves generator and controller.
  2. Self manufactured device inserted into the vaginal cavity and creating subsound pressure waves.
  Arms: Miniature Actilady device active
Device: Miniature Actilady device not active — Devices: Targeted pressure waves are created by two kind of methods ActiLady).
  The effect of the waves used will be examined by the use of a silicon tube or polyvinyl chloride (PVC) tube which is inserted into the vaginal cavity. The other end of the tube will be connected to an "off the shelf" pressure waves generator and controller.
  Self manufactured device inserted into the vaginal cavity and creating subsound pressure waves.
  Arms: Miniature Actilady device not active

SUMMARY:
ActiLady refers is employing targeted pressure waves, with the goal of reducing the pain associated with menstruation (clinically known as dysmenorrhea).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-35 years
2. Regular menstrual cycles (26-35 days); average duration of menstruation ≥5 days for the 4 months preceding the beginning of the trial.
3. Dysmenorrhea pain score >50mm on a 100mm visual analog scale (VAS) for the maximum abdominal pain
4. Analgesic use during every menstrual cycle
5. Non-pregnant, with no intentions to get pregnant during the clinical trial
6. Agrees not to use oral contraceptives or an intrauterine device (IUD) during the trial period
7. Agrees not to use analgesics, except during permitted period (16:00-04:00 the next day, daily)
8. Consents to the use of pads or other vaginal devices throughout the trial period
9. Subject is able to comply with all the requirements of the study and agrees to participate in all the activities of the study
10. Signed written informed consent form (ICF) to participate in the study

Exclusion Criteria:

1. Pregnant or lactating women
2. Used hormonal and/or oral contraceptives in the preceding 4 months
3. Use of an IUD in the preceding 4 months
4. Previous diagnosis of secondary dysmenorrhea
5. Urinary incontinence
6. Duration of menstruation is <5 days
7. Subjects with a known sensitivity to mechanical vibrations and/or silicone
8. Participation in current or recent clinical trial within 30 days prior to baseline visit

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a novel method and device called ActiLady. | 6 months

SECONDARY OUTCOMES:
* Evaluate the pain-reducing effect of ActiLady on dysmenorrhea. * Study the relationship between menses flux and dysmenorrhea. [Time Frame: 6 months] [Designated as safety issue: No ] * Optimize treatment procedure and wave form. | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Hadassah Medical Organization, Jerusalem